CLINICAL TRIAL: NCT04326504
Title: Dolutegravir and Clinical Outcomes Among ART-recipients in Brazil: A Population-based Study
Brief Title: Dolutegravir and Clinical Outcomes Among ART-recipients in Brazil
Acronym: CODE
Status: Recruiting | Type: Observational
Sponsor: Fundação Bahiana de Infectologia (Other)
Collaborators: University of New Mexico (Other); Instituto Infectologia Evandro Chagas, Rio de Janeiro (Unknown); Fundação de Medicina Tropical de Manaus (Unknown); Hospital de Clinicas de Porto Alegre (Other); Centro de Referência e Tratamento, CRT, São Paulo, SP (Unknown); Hospital Partenon, Porto Alegre (Unknown); Universidade Municipal de São Caetano do Sul (Unknown); Universidade Federal do Rio Grande do Norte (Other); Hospital Universitário Cassiano Antônio de Moraes/HUCAM (Unknown); Hospital das Clínicas da Faculdade de Medicina de Ribeirao Preto/USP (Unknown); Faculdade de Medicina de Botucatu, Unesp (Unknown); Sociedade Campineira de Educação e Instrução - Campinas (Unknown); Fundação Universidade de Caxias do Sul - FUCS/RS (Unknown)
Responsible Party: Sponsor
Other Study IDs: FBAI
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections; Clinical Outcomes; Adverse Drug Event; Effect of Drugs
MeSH Terms: conditions — HIV Infections; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients starting DTG-based regimens: ART-naïve patients, starting cART regimens based on DTG
  Interventions: Other: No intervention
- Switch cohort: Patients on stable ART regimens switching to DTG (any reason)
  Interventions: Other: No intervention
- Therapy failure: ART-experienced patients switching to DTG-containing regimens due to virological failure
  Interventions: Other: No intervention
- Non-DTG group: Patients who started a non-DTG containing regimen
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This will be an observational study, no intervention will be performed

SUMMARY:
Access to antiretroviral therapy (ART) in low-income and middle-income countries has been scaled-up effectively over recent years. Recently, the World Health Organization (WHO) guidelines changed to recommend the use of Dolutegravir (DTG) combined with two nucleoside reverse transcriptase inhibitors (NRTIs), tenofovir and lamivudine, for first-line ART; however, there is still a need for further data on the outcomes of DTG-based regimens for people with HIV-1.

This study aims to describe the outcomes of drug-naïve and experienced patients starting a dolutegravir (DTG)-based regimen in a large cohort of HIV - infected patients in Brazil and compare to outcomes obtained from a retrospective control group of subjects who initiated non-DTG-based ART.

DETAILED DESCRIPTION:
CODE is a multicenter prospective observational study to describe and quantify the outcomes of patients starting DTG-based regimens. The investigators will follow ART-naïve patients starting DTG-based regimens (Group 1), patients on stable ART regimens switching to DTG (any reason) (Group 2), and ART-experienced patients switching to DTG-containing regimens due to virological failure (Group 3). In addition, for comparison purposes, the investigators will collect data on patients who started a non-DTG containing regimen (Group 4) in the period for 2014-2016 and did not switch to DTG-based regimens (Figure 1). Enrolled patients will be followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent.

  * HIV infection documented by plasma HIV RNA viral load, a rapid HIV test or any licensed ELISA test; and confirmed by another test using a different method, including but not limited to a rapid HIV test, Western Blot, HIV culture, HIV antigen, or HIV pro-viral DNA at any time prior to study entry.
  * Age ≥ 15 years.
  * For women of child-bearing potential, willingness to use effective contraceptives.
  * Starting use of DTG-based regimen, or being initiated on a non-DTG based ART between 2014 - 2016.

Exclusion Criteria:

* • Any previous use of ART (drug-naïve group only).

  * Current imprisonment, or compulsory detention (involuntary incarceration). For treatment of a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CODE is a multicenter prospective observational study to describe and quantify the outcomes of patients starting DTG-based regimens. The investigators will follow ART-naïve patients starting DTG-based regimens (Group 1), patients on stable ART regimens switching to DTG (any reason) (Group 2), and ART-experienced patients switching to DTG-containing regimens due to virological failure (Group 3). In addition, for comparison purposes, the investigators will collect data on patients who started a non-DTG containing regimen (Group 4) in the period for 2014-2016 and did not switch to DTG-based regimens (Figure 1).
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
frequency of therapy discontinuation due to any event for patients starting ART | 36 months
  The key outcomes of interest include treatment discontinuation due to any event as well as specifically due to metabolic and psychiatric events, virologic outcomes (viral suppression at 12 months, failure to ART, and genotypic results of acquired resistance), clinical outcomes (including noted side effects, retention in care, death, weight changes, hyperglycemia, diabetes, lipid changes, AIDS-defining illnesses, and recorded psychiatric and CNS effects), and special outcomes / populations (pregnancy outcomes, IRIS events, changes in HRQoL, viral hepatitis flares, and tuberculosis outcomes)
therapy discontinuation due to any event for ART-eprerienced patients starting DTG-based regimens | 36 months
  therapy discontinuation due to any event for ART-experienced patients

SECONDARY OUTCOMES:
Exploratory outcomes | 36 months
  These clinical outcomes include: all-cause mortality; all AIDS-defining events; all types of cancer; bacterial pneumonia; pulmonary embolism; deep vein thrombosis; new-onset diabetes mellitus (as defined by the ADA criteria);10 coronary artery disease requiring drug treatment; congestive heart failure; peripheral vascular disease; fractures; and solicited adverse events.
Changes in quality of life for patients switching to DTG-based regimens | 6 and 12 months
  Physical and Mental Components Scores will be measured. HRQoL evaluation will be performed only for patients switching to DTG-based regimens, at the time switch occurs (baseline), and after 6 and 12 months of follow up.
HIV drug resistance | 36 months
  This outcome will be evaluated by collecting samples of blood prior to starting DTG-based ART. These tests will not be done in real time, and results will not be given to the investigator or participant. Once virological failure is identified, the baseline sample will be used to assess transmitted drug resistance through comparison with current resistance genotypic tests. Key mutations that are associated with viral resistance will be determined using information periodically updated by the International AIDS Society.
Markers of CVD risk | 36 months
  Assessments will be made of blood lipids, smoking, blood pressure, incidence of diabetes mellitus, use of medication to lower blood pressure and lipids, and the use of aspirin, to assist in the evaluation of cardiovascular risks and benefits of early treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Fundação Bahiana de Infectologia/SEI, Salvador, Estado de Bahia
  - Fundação Bahiana de Infectologia, Salvador, Estado de Bahia
  - Centro de Referência e Treinamento, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dutertre M, Cuzin L, Demonchy E, Pugliese P, Joly V, Valantin MA, Cotte L, Huleux T, Delobel P, Martin-Blondel G; Dat'AIDS Study Group. Initiation of Antiretroviral Therapy Containing Integrase Inhibitors Increases the Risk of IRIS Requiring Hospitalization. J Acquir Immune Defic Syndr. 2017 Sep 1;76(1):e23-e26. doi: 10.1097/QAI.0000000000001397. No abstract available. PMID 28418992
- [Result] de Boer MG, van den Berk GE, van Holten N, Oryszcyn JE, Dorama W, Moha DA, Brinkman K. Intolerance of dolutegravir-containing combination antiretroviral therapy regimens in real-life clinical practice. AIDS. 2016 Nov 28;30(18):2831-2834. doi: 10.1097/QAD.0000000000001279. PMID 27824625
- [Result] Ciccullo A, Baldin G, Cossu MV, Passerini M, Borghetti A, Capetti A, Di Giambenedetto S. Dolutegravir Plus Lamivudine as First-Line Regimen in a Multicenter Cohort of HIV-1-Infected Patients: Preliminary Data from Clinical Practice. AIDS Res Hum Retroviruses. 2020 Jan;36(1):4-5. doi: 10.1089/AID.2019.0147. Epub 2019 Sep 30. No abstract available. PMID 31476877
- [Result] Elzi L, Erb S, Furrer H, Cavassini M, Calmy A, Vernazza P, Gunthard H, Bernasconi E, Battegay M; Swiss HIV Cohort Study Group. Adverse events of raltegravir and dolutegravir. AIDS. 2017 Aug 24;31(13):1853-1858. doi: 10.1097/QAD.0000000000001590. PMID 28692533
- [Result] Hoffmann C, Welz T, Sabranski M, Kolb M, Wolf E, Stellbrink HJ, Wyen C. Higher rates of neuropsychiatric adverse events leading to dolutegravir discontinuation in women and older patients. HIV Med. 2017 Jan;18(1):56-63. doi: 10.1111/hiv.12468. Epub 2016 Nov 10. PMID 27860104
- [Result] Norwood J, Turner M, Bofill C, Rebeiro P, Shepherd B, Bebawy S, Hulgan T, Raffanti S, Haas DW, Sterling TR, Koethe JR. Brief Report: Weight Gain in Persons With HIV Switched From Efavirenz-Based to Integrase Strand Transfer Inhibitor-Based Regimens. J Acquir Immune Defic Syndr. 2017 Dec 15;76(5):527-531. doi: 10.1097/QAI.0000000000001525. PMID 28825943
- [Result] Taramasso L, Ricci E, Menzaghi B, Orofino G, Passerini S, Madeddu G, Martinelli CV, De Socio GV, Squillace N, Rusconi S, Bonfanti P, Di Biagio A; CISAI Study Group. Weight Gain: A Possible Side Effect of All Antiretrovirals. Open Forum Infect Dis. 2017 Nov 3;4(4):ofx239. doi: 10.1093/ofid/ofx239. eCollection 2017 Fall. PMID 29255735
- [Result] Zash R, Makhema J, Shapiro RL. Neural-Tube Defects with Dolutegravir Treatment from the Time of Conception. N Engl J Med. 2018 Sep 6;379(10):979-981. doi: 10.1056/NEJMc1807653. Epub 2018 Jul 24. No abstract available. PMID 30037297
- [Result] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228
- [Result] Cruz LN, Fleck MP, Oliveira MR, Camey SA, Hoffmann JF, Bagattini AM, Polanczyk CA. Health-related quality of life in Brazil: normative data for the SF-36 in a general population sample in the south of the country. Cien Saude Colet. 2013 Jul;18(7):1911-21. doi: 10.1590/s1413-81232013000700006. PMID 23827895
- [Result] Laguardia J, Campos MR, Travassos C, Najar AL, Anjos LA, Vasconcellos MM. Brazilian normative data for the Short Form 36 questionnaire, version 2. Rev Bras Epidemiol. 2013 Dec;16(4):889-97. doi: 10.1590/s1415-790x2013000400009. English, Portuguese. PMID 24896594